CLINICAL TRIAL: NCT02489006
Title: A Phase II, Open-Label, Randomized, Multi-Centre Study, of Neoadjuvant Olaparib in Patients With Platinum Sensitive Recurrent High Grade Serous Ovarian/Primary Peritoneal or Fallopian Tube Cancer
Brief Title: A Study of Olaparib Prior to Surgery and Chemotherapy in Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Acronym: NEO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZM-058
Record Dates: First submitted 2015-04-17; First posted 2015-07-02 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Neoadjuvant Treatment; Debulking Surgical Procedures
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — olaparib; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olaparib Prior to Surgery, Chemotherapy/Olaparib Post Surgery (Experimental): Olaparib, orally, at 300 mg twice per day, for 6 weeks (+/- 2 weeks) prior to surgery.
  Platinum-based chemotherapy chosen by the study doctor and per standard of care after surgery.
  Olaparib, orally, at 300 mg twice per day, continuously, after chemotherapy.
  Interventions: Drug: Olaparib; Drug: Platinum-based Chemotherapy
- Olaparib Prior to Surgery and Post Surgery (Experimental): Olaparib, orally, at 300 mg twice per day, for 6 weeks (+/- 2 weeks) prior to surgery and after surgery.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib
  Other Names: Lynparza
Drug: Platinum-based Chemotherapy — Chosen by the study doctor, per standard of care.
  Arms: Olaparib Prior to Surgery, Chemotherapy/Olaparib Post Surgery

SUMMARY:
This is a study that will look at the effects and how useful investigational drug olaparib is as a neoadjuvant treatment (treatment given as to shrink a tumor before the main treatment) prior to surgery in patients with recurrent ovarian, primary peritoneal or fallopian tube cancer.

DETAILED DESCRIPTION:
Olaparib belongs to a class of anti-cancer agents known as poly ADP-ribose polymerase (PARP) inhibitors. Olaparib is a new type of drug for ovarian cancer. Laboratory tests show that it may help slow the growth of ovarian cancer.

Olaparib works by blocking the PARP protein. PARP is an important protein which tries to fix damaged deoxyribonucleic acid (DNA, molecules that contain important instructions for the development of cells). Many cancers are thought to develop from damaged DNA. Research has shown that PARP inhibitors stop the PARP protein from working, and that sometimes that can cause cancer cells to stop growing or die.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent high grade serous ovarian/primary peritoneal or fallopian tube cancer.
* Patients must have disease amenable to pre-operative biopsy.
* Patients must have disease deemed suitable for surgical debulking.
* Patients must have a progression free interval of at least 6 months prior to registration.
* Patients must have had at least one line of platinum based therapy.
* Patients must have shown platinum sensitivity to their last line of platinum therapy
* Age >=18 years
* ECOG performance status 0-1 within 7 days of registration
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function
* Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.
* Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib.
* History of allergic reactions attributed to platinum precluding further use.
* Radiation therapy within 4 weeks of registration
* Use of any other systemic, targeted, immunotherapy, chemotherapy, or investigational agents within 4 weeks of registration
* Previously received a PARP inhibitor
* Other malignancy within the last 2 years with exceptions
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Concomitant use of known potent CYP3A4 inhibitors
* Concomitant use of known potent CYP3A4 inducers
* Other anti-cancer therapy including immunotherapy, hormonal therapy, biological therapy, other novel agents or investigational agents
* Persistent toxicities (CTCAE v 4.03 grade >2) caused by previous cancer therapy, excluding alopecia
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Patients with brain metastases
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Patients with known active hepatitis (i.e., hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Pregnant or breastfeeding women
* Receipt of live attenuated vaccine within 30 days prior to enrollment
* Patients with > Grade 2 hearing impairment as per CTCAE v 4.03
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2016-07-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in levels of PAR or PARP-1 before and after study treatment | 4-8 weeks
Mutations in BRCA1/2, RAD51B, RAD51C, RAD51D, PPM1D, FANCM, BRIP1, PALB2 and BARD1 in germline tissue compared to tumor tissue | 2.5 years

SECONDARY OUTCOMES:
Frequency of adverse events, by description and grade | 2.5 years
Response rate to olaparib in the neoadjuvant period | 6 weeks
Duration of progression free survival with olaparib in comparison to platinum based chemotherapy | 2.5 years
Levels of ctDNA compared to levels of CA125 | 2.5 years
Gene expression changes in tumour tissue before and after treatment with Olaparib | 2.5 years
Secondary mutation rate in surgical tumour specimens following PARP therapy and at progression | 2.5 years
  2.5 years
Changes in blood based biomarkers using ctDNA before, during and after treatment with Olaparib | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (9):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Vall d'Hebron University Hospital, Barcelona, Spain
- United Kingdom (2):
  - Royal Marsden Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London